CLINICAL TRIAL: NCT00604916
Title: The Effectiveness of an Oral Care Protocol in Preventing Ventilator- Associated Pneumonia for Intensive Care Unit Patient
Brief Title: Oral Care Protocol for Preventing Ventilator- Associated Pneumonia
Acronym: VAP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Collaborators: National Taiwan University (Other)
Responsible Party: li-yin YAO, School of Nursing, National Taiwan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MMH-I-S-402
Record Dates: First submitted 2008-01-07; First posted 2008-01-30 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2008-01

CONDITIONS: Pneumonia
Keywords: oral hygiene
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- E (Experimental): received a 7 day standardized oral care protocol
  Interventions: Other: standardized oral care protocol - electronic toothbrush
- C (Placebo Comparator): received a 7 day mimic protocol
  Interventions: Other: mimic protocol

INTERVENTIONS:
Other: standardized oral care protocol - electronic toothbrush — a standardized 20-minute oral care protocol using an electronic toothbrush to clean and moisturize oral cavity twice daily.
  Arms: E
Other: mimic protocol — a mimic 20-minute protocol involving moisturizing and attention control was performed for the same intervals.
  Arms: C

SUMMARY:
The Nosocomial Pneumonia remains to be a major complication for patients who were incubated with ventilation. Most cases are attributed to increased bacteria flora in oropharyngeal secretion and aspiration of those organisms. Research indicates that the Gram-Negative Bacteria grows in upper air way and trachea rapidly during the initial 2-4 hospital days and the dental plague also increased dramatically at the first 5 days. About 50% cases with prolonged intubation experienced temporal swallowing disorders and majority of them recovered 7 days post weaning. Some evidence exist suggesting that oral care could reduce bacterial flora, prevent aspiration, and subsequently decrease the incidence of ventilation-associated pneumonia for this group of high risk patients.

This study aims to evaluate the effectiveness of a standardized oral care protocol in improving oral hygiene and reducing the incidence of pneumonia on a sample of surgical patients at intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly admitted to SICU who were under ventilator support for 48~72 hours

Exclusion Criteria:

* With pneumonia present

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-03; Primary Completion 2007-11 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
the oral hygiene status measured by the oral assessment guide and plague index | every 3~4days

SECONDARY OUTCOMES:
The incidence of VAP defined by the Clinical Pulmonary Infection Score | a 7 day oral care protocol duration

CONTACTS AND LOCATIONS:
Overall Officials: li-yin YAO, BSN, Principal Investigator — School of Nursing, National Taiwan University